CLINICAL TRIAL: NCT02413658
Title: Phenytoin in the Healing of Clean Surgical Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Surgical Center, Cambodia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1CSC2015
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Wound; Re-Epithelialization
Keywords: Phenytoin; Skin graft donor site; Clean surgical site; Wound model
MeSH Terms: conditions — Wounds and Injuries | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Control (Active Comparator): Dressings of best current clinical practice, sugar solution.
  Interventions: Drug: Sugar solution
- Phenytoin 1 (Experimental): Dressings using phenytoin solution 20mg/ml
  Interventions: Drug: Phenytoin
- Phenytoin 2 (Experimental): Dressings using phenytoin solution 40mg/ml
  Interventions: Drug: Phenytoin

INTERVENTIONS:
Drug: Phenytoin — Topical use of phenytoin solution on dressings of split thickness skin graft sites.
  Other Names: Dilantin, Dilantin-125
  Arms: Phenytoin 1; Phenytoin 2
Drug: Sugar solution
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the potential healing properties of phenytoin.

The investigators will use the donor site of a split skin thickness graft (SSTG) to model a basic wound in a randomized controlled trial of topical phenytoin against current best clinical practice. The investigators aim to demonstrate a dose dependent effect. The investigators hypothesis, based on previous clinical experience at our center and on current available literature, that phenytoin will reduce wound healing time.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing split thickness skin graft during trial time period at Children's Surgical Centre

Exclusion Criteria:

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Percentage rate of re-epithelialization | Participants will be followed for the duration of hospital stay, an expected average of 20 days
  Pictures taken of wound site every other day will be analysed using imaging software for size of wound. Percentage rate will be calculated from this.
Appearance of infection | Participants will be followed for the duration of hospital stay, an expected average of 20 days
  Pictures taken of wound site every other day will be analysed using imaging software and the Southampton wound grading scale

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Surgical Centre, Phnom Penh, Cambodia